CLINICAL TRIAL: NCT04611633
Title: A Prospective Observational Study in COPD Patients Evaluating the Quality of Life in Patients Switching From a Dual Therapy to a Fixed LABA/LAMA/ICS Triple Therapy in Routine Practice
Brief Title: Study in COPD Patients Evaluating the Quality of Life (TRISNOOZE)
Acronym: TRISNOOZE
Status: Terminated | Type: Observational
Why Stopped: Due to COVID pandemic not feasible to include patients for this study
Sponsor: Chiesi SA/NV (Other)
Responsible Party: Sponsor
Other Study IDs: CHIESI_NIS_004
Record Dates: First submitted 2020-10-27; First posted 2020-11-02 (Actual); Last update posted 2021-12-09 (Actual); Status verified 2021-11

CONDITIONS: Chronic Obstructive Pulmonary Disease
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Combination Product: Trimbow — As this is a non-interventional study, all treatment decisions will be made at the discretion of the treating physician prior to enrolment in the study and during the entire period of the study. Treatment will be prescribed according to the product label in the summary of product characteristics.

SUMMARY:
This non-interventional study aims to collect information on the patient's quality of life, as well as the quality of sleep when stepping up to a fixed triple maintenance therapy (Trimbow®) as per physicians' decision, independent from study participation, and to assess its effectiveness in daily life, in general practitioner setting.

DETAILED DESCRIPTION:
This non-interventional study assesses the real-life effectiveness, with focus on patient's quality of life, of the fixed triple therapy Trimbow® after stepping up from a dual therapy in clinical practice at first line centres in patients with confirmed chronic obstructive pulmonary disease (COPD). Data will be collected on availability as per usual care at baseline, 3 and 6 months after inclusion.

ELIGIBILITY:
Inclusion Criteria:

* Patient has provided written informed consent
* Patient is aged 40 years or older
* Current or ex-smokers with a smoking history ≥ 10 pack years
* Patient is diagnosed with COPD, confirmed by post-bronchodilator spirometry (Tiffeneau index <0.7; baseline or older spirometry)
* Patient is eligible for switch to triple therapy with at least 12 weeks of stable double inhalation therapy (ICS/LABA or LABA/LAMA) prior to enrolment to the study
* Patient is starting treatment with Trimbow® upon decision by their physician

Exclusion Criteria:

* Patients who are hypersensitive to one of the active substances or excipients
* Patients who are treated with triple therapy (via single or multiple inhalers) in the last 6 months prior to study enrolment
* Patients on ICS, LABA or LAMA monotherapy
* Patients with pneumonia and/or a moderate or severe COPD exacerbation not resolved ≥ 14 days prior to screening and ≥ 30 days following the last dose of oral/systemic corticosteroid (if applicable), or a respiratory tract infection not resolved ≥ 7 days prior to screening
* Patients participating simultaneously to other clinical trials or studies

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The subject population will include adult patients aged 40 years or above diagnosed with COPD confirmed by spirometry (Tiffeneau index <0.7), who are stepping up from dual therapy (ICS/LABA or LABA/LAMA treatment at least 12 weeks prior to enrolment to the study) to a fixed triple maintenance therapy (Trimbow).
  Approximately 800 patients are expected to be enrolled at 200 GP practices in Belgium.
Sampling Method: Probability Sample
Enrollment: 14 (Actual)
Dates: Start 2021-01-18 (Actual); Primary Completion 2021-09-16 (Actual); Study Completion 2021-09-16 (Actual)

PRIMARY OUTCOMES:
COPD symptoms | 6 months
  The patient's COPD symptoms at month 6 (visit 3), compared to baseline. This is measured by the COPD Assessment Test (CAT) questionnaire.

SECONDARY OUTCOMES:
COPD symptoms | 3 months
  The patient's COPD symptoms at month 3 (visit 2)
Quality of sleep | 6 months
  The quality of sleep of the patients using the CASIS questionnaire at baseline, month 3 and 6 (visit 2 and 3)
Treatment satisfaction | 6 months
  The patient's treatment satisfaction score using PGI-C at month 3 and 6 (visit 2 and 3)
Rescue medication | 6 months
  Use of rescue medication at baseline and each follow-up visit (question on the past 7 days)
Lung function parameters | 6 months
  Lung function parameters (FEV1, FVC) (if available) at baseline and each follow-up visit

OTHER OUTCOMES:
Moderate/severe exacerbations | 6 months
  Number of moderate/severe exacerbations at baseline and at month 6

CONTACTS AND LOCATIONS:
Overall Officials: Eric Marchand, MD, PhD, Principal Investigator — CHU Godinne UCL Namur
Locations (11):
- Belgium (11):
  - General practitioners in the province of East Flanders, Ghent, East Flanders
  - General practitioners in the province of Flemish Brabant, Leuven, Flemish Brabant
  - General practitioners in the province of Hainaut, Mons, Hainaut
  - General practitioners in the province of Limburg, Hasselt, Limburg
  - General practitioners in the province of Luxembourg, Arlon, Luxembourg
  - General practitioners in the province of Walloon Brabant, Wavre, Walloon Brabant
  - General practitioners in the province of West Flanders, Bruges, West Flanders
  - General practitioners in the province of Antwerp, Antwerp
  - General practitioners in the province of Liège, Liège
  - CHU-UCL-Namur, Namur
  - General practitioners in the province of Namur, Namur